CLINICAL TRIAL: NCT02918435
Title: Implementing an Intervention to Address Social Determinants of Health in Pediatric Practices
Acronym: PROSWECARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Pediatric Research in Office Settings (Network); Continuity Research Network (Network); Boston University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Arvin Garg, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: H-35482; R01HD090191 (NIH)
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Basic Unmet Material Needs; Patient Satisfaction; Receipt of Community Resources; Provider Referrals
Keywords: WE CARE; Pediatric practices
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care-Control (No Intervention): Participants in the usual care group will receive standard pediatric care.
- On-site WE CARE implementation arm (Experimental): WE CARE will be implemented in the study site using a facilitated "on-site" strategy. 1. Participants will receive the WE CARE survey at health supervision visits; this survey will be used to identify unmet material needs. 2. Providers will be trained on WE CARE via an on-site team which will teach them how to review the survey and provide referrals (community resource information sheets) from a Family Resource Book located in each exam room.
  Interventions: Behavioral: WE CARE
- Self-directed web-based WE CARE implementation arm (Experimental): WE CARE will be implemented in the study site using a web-based implementation strategy. 1. Participants will receive the WE CARE survey at health supervision visits; this survey will be used to identify unmet material needs. 2. Providers will be trained on WE CARE via web-based tools (e.g., web-based seminar) which will teach them how to review the survey and provide referrals (community resource information sheets) from a Family Resource Book located in each exam room
  Interventions: Behavioral: WE CARE

INTERVENTIONS:
Behavioral: WE CARE — The WE CARE (Well-child care visit, Evaluation, Community Resources, Advocacy, Referral, Education) survey consists of 12 questions used to identify six unmet material needs (education, employment, food security, housing, childcare, household utilities). It will be administered at health supervision visits during the WE CARE phase at each study site. The Family Resource Book will contain resource information sheets for each of these needs listing available community resources. A physician champion will conduct regular booster sessions every 4 months and train new providers should there be staff turnover.
  Arms: On-site WE CARE implementation arm; Self-directed web-based WE CARE implementation arm

SUMMARY:
This research project is aimed to assess the implementation, effectiveness, and sustainability of a pediatric-based intervention aimed at reducing families' unmet material needs (food, housing, employment, childcare, household utilities, education) in pediatric practices throughout the United States.

DETAILED DESCRIPTION:
The investigators prior work has focused on developing a pediatric primary care-based intervention, WE CARE (Well-child care visit, Evaluation, Community Resources, Advocacy, Referral, Education), aimed at addressing poor families' material needs - food security, employment, parental education, housing stability, household heat, and childcare - by systematically screening for these needs and referring families to existing community-based services. To date, the investigators have tested WE CARE primarily in community health centers (CHCs); their randomized controlled trial (RCT) demonstrated WE CARE's efficacy on parental receipt of community-based resources. However, over 80% of low-income children receive care from providers in traditional pediatric practices (i.e. non-CHCs). The investigators therefore will conduct a large-scale, Hybrid Type 2 effectiveness-implementation trial in eighteen pediatric practices in the US. A stepped wedge study cluster RCT design will be used to implement WE CARE in all practices using two common strategies used to integrate systems-based interventions into primary care - a previously facilitated "on-site" strategy in which content experts provide training sessions and on-going consultation; and a self-directed "web-based" method modeled after the American Academy of Pediatrics' practice transformation strategy. The proposed study's specific aims are to: 1) demonstrate the non-inferiority of the self-directed, web-based strategy for implementing WE CARE, in comparison to the facilitated on-site strategy; 2) demonstrate WE CARE's effectiveness on increasing parental receipt of community resources; and 3) assess the sustainability of WE CARE in pediatric practices. The investigators hypothesize that WE CARE will have equivalent fidelity via the two strategies. Based on prior work, the investigators hypothesize that WE CARE will significantly increase parental receipt of community resources three months post-visit compared to usual care. The investigators also expect WE CARE to be sustained 1.5-, 2-, and 2.5-years post-implementation; they expect to gather data from over 2,700 chart reviews, 2,520 parent-child dyads, and 360 providers and office staff. This proposal has significant public health implications for the delivery of primary care to low-income children.

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians (aged at least 18 years) of children aged 2 months through 10 years whose child presents for a health supervision visit

Exclusion Criteria:

* Foster parents, parents who speak neither English or Spanish, and previously enrolled parents

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1872 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Receipt of Community Resources | 3 months post-index visit
  Effectiveness outcome of WE CARE (Well-child care visit, Evaluation, Community Resources, Advocacy, Referral, Education) on parental receipt of community resources
Provider Referrals for Unmet Material Needs at Visit | Baseline at Index visit
  Implementation outcome of WE CARE on provider referrals

SECONDARY OUTCOMES:
WE CARE survey distribution | 1.5-,2-,and 2.5- years post-implementation of WE CARE
  Sustainability of WE CARE- office staff outcome
Appropriate referrals made by providers | 1.5-,2-,and 2.5- years post-implementation of WE CARE
  Sustainability of WE CARE- provider outcome
Patient satisfaction measured via the CAHPS Clinician and Group Survey (Child) | 3 months post-index visit
  Parental assessment of satisfaction of pediatric care received
Family centeredness measured via the National Survey of Children's Health (2016) | 3 months post-index visit
  Parental assessment of family centeredness of pediatric care received
Care coordination measured via the National Survey of Children's Health (2016) | 3 months post-index visit
  Parental assessment of the care coordination of pediatric care received
Acceptability of WE CARE measured via questionnaires | Through study completion; baseline and 12-15 months into WE CARE phase at all sites
  Providers and Office staff acceptability views on WE CARE
Whether Discussion of Unmet Needs (e.g., food insecurity) occurred at child's well-child care visit | Baseline at index visit
  Measurement of whether discussion of unmet social needs occurred during pediatric visit
Appropriateness of WE CARE measured via questionnaire | Through study completion; baseline and 12-15 months into WE CARE phase at all sites
  Providers and Office staff appropriateness views on WE CARE

CONTACTS AND LOCATIONS:
Overall Officials: Arvin Garg, MD, MPH, Principal Investigator — University of Massachusets Medical School
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg A, Toy S, Tripodis Y, Silverstein M, Freeman E. Addressing social determinants of health at well child care visits: a cluster RCT. Pediatrics. 2015 Feb;135(2):e296-304. doi: 10.1542/peds.2014-2888. Epub 2015 Jan 5. PMID 25560448
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Thompson RE, Serwint JR. Improving the management of family psychosocial problems at low-income children's well-child care visits: the WE CARE Project. Pediatrics. 2007 Sep;120(3):547-58. doi: 10.1542/peds.2007-0398. PMID 17766528